CLINICAL TRIAL: NCT03023826
Title: Relative Bioavailability and Food Effect Study in Healthy Subjects Administered Two Different Formulations of LY3202626
Brief Title: A Study of LY3202626 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15567; I7X-MC-LLCE (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-01-16; First posted 2017-01-18 (Estimated); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — LY3202626

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3202626 (R-Fasting) (Experimental): Single oral dose of LY3202626 (R) capsule under fasting conditions.
  Interventions: Drug: LY3202626 (R-Fasting)
- LY3202626 (T1-Fasting) (Experimental): Single oral dose of LY3202626 (T1) tablet under fasting conditions.
  Interventions: Drug: LY3202626 (T1-Fasting)
- LY3202626 (T1-Fed) (Experimental): Single oral dose of LY3202626 (T1) following a high fat breakfast.
  Interventions: Drug: LY3202626 (T1-Fed)

INTERVENTIONS:
Drug: LY3202626 (R-Fasting) — Administered orally
  Arms: LY3202626 (R-Fasting)
Drug: LY3202626 (T1-Fasting) — Administered orally
  Arms: LY3202626 (T1-Fasting)
Drug: LY3202626 (T1-Fed) — Administered orally
  Arms: LY3202626 (T1-Fed)

SUMMARY:
The purposes of this study are to determine:

* If there are any differences in the way LY3202626 is handled by the body when taken in two different forms
* Whether a high fat meal affects the way the body handles LY3202626
* How well tolerated LY3202626 is

There are three (3) study periods for all participants. Participants will be admitted to the clinical research unit (CRU) each period and will be discharged from the CRU following the completion of 2 overnight stays and up to 36 hours after dosing with LY3202626.

The study will last about 50 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Female participants must be of non-childbearing potential confirmed by medical history or menopause
* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per meter squared (kg/m²) inclusive, at screening

Exclusion Criteria:

* Are investigative site personnel directly affiliated with this study and their immediate families
* Are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed
* Have previously completed or withdrawn from this study or any other study investigating LY3202626, and have previously received the investigational product
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Have a history of head trauma with loss of consciousness within the last 5 years
* Have known or ongoing psychiatric disorders

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-15; Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 6 sequences in 3 periods.
Groups:
- Sequence (ACB); Sequence (CAB); Sequence (BAC); Sequence (ABC); Sequence (BCA); Sequence (CBA): A: Reference (R): Single oral 12 milligram (mg) dose of LY3202626 capsule (R) under fasting conditions.
  B: Test (T1-12): Single oral 12 mg dose of LY3202626 tablet (T1) under fasting conditions.
  C: Test (T1-12): Single oral 12 mg dose of LY3202626 tablet (T1) following a high fat breakfast.
Period: Period 1
Arm/Group | Sequence (ACB) | Sequence (CAB) | Sequence (BAC) | Sequence (ABC) | Sequence (BCA) | Sequence (CBA)
Started | 4 | 4 | 5 | 4 | 4 | 5
Received at Least One Dose of Study Drug | 4 | 4 | 5 | 4 | 4 | 5
Completed | 4 | 4 | 5 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence (ACB) | Sequence (CAB) | Sequence (BAC) | Sequence (ABC) | Sequence (BCA) | Sequence (CBA)
Started | 4 | 4 | 5 | 4 | 3 | 5
Completed | 4 | 4 | 5 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence (ACB) | Sequence (CAB) | Sequence (BAC) | Sequence (ABC) | Sequence (BCA) | Sequence (CBA)
Started | 4 | 4 | 5 | 4 | 3 | 5
Completed | 4 | 4 | 5 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: Single oral 12 mg dose of LY3202626 capsule (R) under fasting conditions, LY3202626 tablet (T1) under fasting conditions and LY3202626 tablet (T1) following a high-fat meal.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3202626
Description: Pharmacokinetics (PK) is the maximum observed drug concentration (Cmax) of LY3202626
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168 Hours Postdose
Population: All randomized participants who received at least one dose and who had evaluable PK data.
Measure: Geometric Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Groups:
- 12 mg LY3202626 (R-Fasting): Single oral 12 mg dose of LY3202626 capsule (R) under fasting conditions.
- 12 mg LY3202626 (T1-Fasting): Single oral 12 mg dose of LY3202626 tablet (T1) under fasting conditions.
- 12 mg LY3202626 (T1-Fed): Single oral 12 mg dose of LY3202626 tablet (T1) following a high fat breakfast.
Arm/Group | 12 mg LY3202626 (R-Fasting) | 12 mg LY3202626 (T1-Fasting) | 12 mg LY3202626 (T1-Fed)
Number analyzed (Participants) | 25 | 25 | 25
nanogram/milliliter (ng/mL) | 27.9 (64) | 36.1 (45) | 39.4 (42)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of LY3202626
Description: PK is the area under the concentration versus time curve from time zero to infinity (AUC[0-∞]) of LY3202626
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | 12 mg LY3202626 (R-Fasting) | 12 mg LY3202626 (T1-Fasting) | 12 mg LY3202626 (T1-Fed)
Number analyzed (Participants) | 25 | 24 | 25
hour*nanogram/milliliter (h*ng/mL) | 540 (62) | 707 (45) | 702 (46)

3. Primary Outcome: PK: AUC From Time Zero to Time t, Where t is the Last Time Point With a Measurable Concentration (AUC[0-tlast]) of LY3202626
Description: PK is the AUC from time zero to time t, where t is the last time point with a measurable concentration (AUC[0-tlast]) of LY3202626
Time Frame: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and who had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 12 mg LY3202626 (R-Fasting) | 12 mg LY3202626 (T1-Fasting) | 12 mg LY3202626 (T1-Fed)
Number analyzed (Participants) | 25 | 25 | 25
h*ng/mL | 531 (62) | 667 (47) | 691 (45)

ADVERSE EVENTS:
Time Frame: Baseline to End of Study (Up to 3 Months)
Arm/Group | 12 mg LY3202626 (R-Fasting) | 12 mg LY3202626 (T1-Fasting) | 12 mg LY3202626 (T1-Fed)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 8/25 | 7/26 | 9/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 mg LY3202626 (R-Fasting) (N=25) | 12 mg LY3202626 (T1-Fasting) (N=26) | 12 mg LY3202626 (T1-Fed) (N=25)
Catheter site bruise (General disorders) | 1 (1) | 1 (1) | 3 (3)
Catheter site erythema (General disorders) | 3 (3) | 3 (3) | 2 (2)
Catheter site pruritus (General disorders) | 1 (1) | 1 (1) | 2 (2)
Catheter site swelling (General disorders) | 2 (2) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 4 (4) | 1 (1) | 5 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT03023826/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT03023826/SAP_001.pdf